CLINICAL TRIAL: NCT04093154
Title: VR During Accessing a Port With Huber Needle
Brief Title: Effect of VR on Pain, Fear and Anxiety During Accessing a Port With Huber Needle in Pediatric Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, Asistant Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3481GOA 2017/20-01
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Pain; Fear; Anxiety State
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective, parallel trial design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Standard Care + VR VR applications introduced to the child or adolescent by the researcher before the procedure. Three VR applications were used in this study; riding a rollercoaster (Rilix VR), swimming with marine animals in underwater world (Ocean Rift) and exploring the forest though the eyes of woodland species (In the eyes of animal). Children/adolescent chose one of these three applications. When the child is ready for the procedure, the researcher started the application by wearing virtual glasses to the child/adolescent. VR intervention was started 2-3 min before the procedure and continued until the procedure was completed.
  Interventions: Device: wearing the virtual headset
- Control (No Intervention): Standart Care Control group children did not receive any distraction techniques.

INTERVENTIONS:
Device: wearing the virtual headset — watching the application by wearing virtual glasses to the child/adolescent
  Arms: Virtual Reality

SUMMARY:
Virtual Reality (VR) can be used during needle-related procedures in children with cancer. The aim of this study was to investigate the effect of VR during access the venous port with Huber needle-related pain, fear and anxiety of children and adolescents with cancer.

DETAILED DESCRIPTION:
Study hypotheses H1: The venous port access-related pain, fear and anxiety scores of patients in VR group during access the venous port with Huber needle is lower from the control group.

Methods Study Design and Sample This is a randomized controlled study of virtual reality during access the venous port with Huber needle performed in a pediatric hematology and oncology setting at two university hospital in Izmir. Data were recorded on 42 children and adolescents with cancer aged 6-17 undergoing Huber needle insertion into a subcutaneously implanted intravenous port.

Gpower 3.1.0 statistical program showed that 21 patients in each group were needed based on an effect size of 0.20, at a power of 0.80, and an acceptable type I error size of 0.05.

Randomization Forty-two children enrolled the study. They were allocated by the blocked randomization; gender, age (6-12/13-18), subcutaneously implanted intravenous port insertion time (≤1month/>1month). Randomization was performed with a computerized random-number generator. Forty-six children were assessed for eligibility; 4 children were excluded; refused to participate (n = 2); had visual problem (n = 1); did not want to wear VR glasses to see access the venous port with Huber needle before the procedure (n = 1).

Instruments Demographic Form. This form included the child's gender, age, the last blood draw time, blood draw success and also the parent demographics such as age, educational level.

Wong-Baker FACES (WBS) Pain Rating Scale. This scale uses in children aged 3 and older to rate pain severity, ranges from 0 (very happy/no pain) to 10 (hurts worst).

The Child Fear Scale (CFS). This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear (4).

The Children's Anxiety Meter (CAM-S). The CAM-S assesses children's anxiety and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10).

Procedure The researcher informed the children and their parents about the aim of the study. Children and adolescents with cancer were randomized to either VR or control group. All children underwent standard care in this access the venous port with Huber needle procedure. In standard care: children/adolescents and their parents were informed by the staff at least one hour before the procedure. None pharmacological methods were used in standard care at the accessing the venous port with Huber needle in the units.

CFS and CAM-S were administered by the researcher to the children/adolescent and his/her parent to assess child's fear and anxiety levels about the port needle insertion 5 minutes ago before the procedure. Children/adolescent and his/her parent were blinded to each other score. Parents of children or adolescents were also present during the procedure. All accessing the venous port with Huber needle procedure was performed in patient's room.

Virtual Reality intervention In the VR Group, after the CFS and CAM-S were administered, VR applications introduced to the child or adolescent by the researcher before the procedure. When the child is ready for the procedure, the researcher started the application by wearing virtual glasses to the child/adolescent. VR intervention was started 2-3 min before the procedure and continued until the procedure was completed.

Ethics Ethical approval was received from the Non-Invasive Clinical Studies Ethics Committee of University where the research was conducted (3481GOA 2017/20-01). The researcher informed about the aim of the study and obtained written consent forms from children and parents.

ELIGIBILITY:
Inclusion Criteria:

* aged 6-18 years,
* clinical diagnosis of pediatric cancer,
* had subcutaneously implanted intravenous port ,
* undergoing access the subcutaneously implanted intravenous port with Huber needle.

Exclusion Criteria:

* aged <6 and >18 years,
* septic, dehydrated, vomiting, sedated, medically unstable,
* previously known severe needle insertion phobia,
* no Huber needle had ever inserted before
* reported pain for another reason in the time of access the venous port with Huber needle,
* had cognitive impairment, or visual problem
* children and parents that do not understand and speak Turkish

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | an average of 1 year
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Fear assesed by Child Fear Scale | an average of 1 year
  The Child Fear Scale used. This scale is a one-item self-report measure for measuring pain-related fear in children. This one-item scale consists of five sex-neutral faces. This rating scale ranges from 0 to 4.It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right (4). The rater responds indicates the level of fear. It can be used by the parents and researchers before and during the procedure for children aged 5-10 years.
Anxiety assesed by Children Anxiety Meter-State | an average of 1 year
  It assesses children's anxiety in clinical settings and uses before medical procedures. The CAM is drawn like a thermometer with a bulb at the bottom, also includes horizontal lines at intervals going up to the top. Children are asked to mark how he/she feel "right now" to measure state anxiety. This scale ranges from 0 to 10. Higher values represent higher anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, Study Director — Dokuz Eylul University Nursing Faculty Pediatric Nursing Department
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerceker GO, Bektas M, Aydinok Y, Oren H, Ellidokuz H, Olgun N. The effect of virtual reality on pain, fear, and anxiety during access of a port with huber needle in pediatric hematology-oncology patients: Randomized controlled trial. Eur J Oncol Nurs. 2021 Feb;50:101886. doi: 10.1016/j.ejon.2020.101886. Epub 2020 Dec 1. PMID 33321461